CLINICAL TRIAL: NCT05294744
Title: Utility of the Use of N-acetylcysteine Associated With Conventional Treatment in Patients With Severe Acute Alcoholic Hepatitis (Maddrey> 32)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bioaraba Health Research Institute (Network)
Responsible Party: Principal Investigator, Ana Belén Fernández Laso, Principal Investigator, Bioaraba Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CONACHAA; 2020-004549-35 (EudraCT Number)
Record Dates: First submitted 2021-07-14; First posted 2022-03-24 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Alcoholic Hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Clinical, randomized, controlled, multicenter, parallel and open trial.
Masking Description: This is an open trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corticosteroids (Active Comparator): Corticosteroids following Standard Clinical Practice
  Interventions: Drug: N-acetylcysteine
- Corticosteroids + N-acetylcysteine (Experimental): Corticosteroids following Standard Clinical Practice plus N-acetylcisteine
  Interventions: Drug: N-acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine — Day 1: 150 mg/kg in 250ml 5% glucose over 30min + 50mgr/kg in 500ml glucose over 4h + 100mgr/kg in 1000ml glucose over 16h intravenously.
  Day 2-14: 100mgr/kg in 1000 ml glucose/24h intravenously. Day 15 until end of corticosteroid treatment: NAC 600mg orally every 24h.

SUMMARY:
This study is designed to evaluate the hypothesis that patients with severe acute alcoholic hepatitis have lower morbi-mortality if the patients receive treatment with corticosteroids + NAC, compared to patients that only receive corticosteroids.

DETAILED DESCRIPTION:
Currently there are no drugs available to cure patients with acute alcoholic hepatitis. The only treatment available is corticosteroids, the efficacy of which is limited and not free of side effects.

Other drugs that can contribute to improve the situation of patients with this entity is N-acetylcysteine (NAC), however, in the different studies contradictory data are obtained, therefore, different societies recommend conducting studies of greater scope to confirm the effectiveness of N-acetylcysteine and to be able to make a clear indication about N-acetylcysteines use.

Clinical, randomized, controlled, multicenter, parallel and open trial.

ELIGIBILITY:
Inclusion Criteria:

* Men and women.
* Age from 18 to 75 years.
* Patients with acute alcoholic hepatitis according to AASLD criteria or compatible liver histology.
* Maddrey score> = 32.
* Acceptance of participation through written informed consent.

Exclusion Criteria:

* Any cause of jaundice: acute hepatitis, positive HIV serology, biliary-pancreatic pathology, hemolytic anemia.
* Allergy or intolerance to N-acetylcysteine and / or corticosteroids.
* Hepatocarcinoma.
* Portal cavernomatosis.
* Portal cavernomatosis.
* Any disease whose life expectancy is less than 12 months.
* Patients with nitroglycerin and / or carbamazepine-based treatments.
* Patients with uncontrolled active infection.
* Acute kidney disease with creatinine> 2.5 mg / dL.
* Uncontrolled upper gastrointestinal bleeding.
* Concomitant uncontrolled diseases (HBV, HCV, HIV, TB, DILI, HCC or acute pancreatitis).
* Multiple organ failure or shock.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2022-10-07 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with all-cause mortality at 6 months. | 6 months.
  Main result variable.

SECONDARY OUTCOMES:
Number of participants with complications: infections, ascites, gastrointestinal bleeding, renal failure, hepatic encephalopathy, need for MARSH or orthotopic liver transplantation. | 3 months
  Security variable.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Belén Fernández, Clinic, Principal Investigator — HUA
Locations (1):
- Ana Belén Fernández Laso, Vitoria-Gasteiz, Álava, Spain

IPD SHARING:
Plan to Share IPD: No
There is no a plan to make individual participant data (IPD) available to other researchers.